CLINICAL TRIAL: NCT03324711
Title: Psychometric Validation of the "Antillanisée" Version of the Mini Mental State Examination
Brief Title: Psychometric Validation of the "Antillanisée" Version of the Mini Mental State Examination (MMSEa)
Acronym: MMENSEA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the Principal Investigator
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15/B/26
Record Dates: First submitted 2017-01-11; First posted 2017-10-30 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Elderly Patients; Cognitive Disorder; Alzheimer Disease
Keywords: Cognitive disorders; Alzheimer's disease; Mini Mental State Examination; Geriatry
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elderly patient (65 and more) (Other): Ederly patients seen in geriatric day hospital, from creole culture.
  Interventions: Diagnostic Test: "Antillanisée" Mini Mental State Examination (MMSEa)

INTERVENTIONS:
Diagnostic Test: "Antillanisée" Mini Mental State Examination (MMSEa) — "Antillanisée" version of the Mini Mental State Examination (MMSEa), is a version adaptated to the French West Indies creole culture.
  Other Names: MMSEa

SUMMARY:
The main objective of the study is to analyze the psychometric properties of the "antillanisée" version of the Mini Mental State Examination (MMSEa).

The methodology used will permit to explore the feasibility, acceptability, validity and reliability of the tool.

The psychometric validation of a version adapted transculturally will increase the value of the results obtained with this test and will make it possible to refine the screening of existing cognitive disorders for elderly subjects with Alzheiner's disease or related disorders.

DETAILED DESCRIPTION:
Patients will be recruited at the Geriatric Day Hospital.

These patients came to a geriatric day hospital for examination without restriction on the reason for the hospitalization.

They are referred by their general practitionner or referred by a specialist physician, live at home or in an institution and are representative of the geriatric population addressed by the MMSEa.

* The main objective of the study is to analyze the psychometric properties of the "antillanisée" version of the Mini Mental State Examination (MMSEa).
* The ancillary objective of this study will be to carry out the psychometric validation of the Short Physical Performance Battery (SPPB) in people aged 65 years or older.

It is an instrument for measuring the physical performance of subjects whose transcultural adaptation and psychometric validation have already been performed in subjects aged 65 to 74 years.

SPPB is used routinely in our routine practice in a day hospital, with no psychometric validation performed on this population. This ancillary objective will not modify the course of the MMSEa validation study since the SPPB is part of the evaluation tools.

ELIGIBILITY:
Inclusion Criteria:

* Subject of 65 years old and over
* Subject admitted in a geriatric day hospital
* Patients of creole culture
* Subject having French and/or Creole as mother tongue
* Subject able to undergo neuropsychological tests
* Subject having given informed consent or, informed consent given by his or her primary caregiver
* Subject affiliated to a social security scheme

Exclusion Criteria:

* Subject with a disability seriously compromising oral communication (understanding and expression)
* Subject with behavioral disorder that does not allow for testing
* Subject in general condition not allowing its participation in the tests
* Subject involved in another study including an exclusion period still in progress at the time of inclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the psychometric properties of the questionnaire MMSEa | 12 month (+/- 15 days)
  The following will be measured:
  * feasibility and acceptability;
  * validity of structure;
  * discriminant validity;
  * predictive validity;
  * validity of convergence;
  * reliability (internal consistency,reproducibility (test-retest)).

SECONDARY OUTCOMES:
Evaluation of the psychometric properties of questionnaire SPPB | 12 month (+/- 15 days)
  The following will be measured:
  * feasibility and acceptability;
  * validity of structure;
  * discriminant validity;
  * predictive validity;
  * reliability (internal consistency,reproducibility (test-retest)).

CONTACTS AND LOCATIONS:
Overall Officials: Lidvine GODAERT-SIMON, MD, Principal Investigator — CHU of Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique, France